CLINICAL TRIAL: NCT06687486
Title: Effect of Autogenic Relaxation Therapy on Caregivers on Perceived Stress Quality of Life and Caregiver Burden: a Randomized Controlled Study
Brief Title: Effect of Autogenic Relaxation Therapy on Caregivers on Perceived Stress Quality of Life and Caregiver Burden
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seda KARAKAYA ERGUN (Other)
Responsible Party: Sponsor-Investigator, Seda KARAKAYA ERGUN, Principal Investigator, Necmettin Erbakan University
Organization: Necmettin Erbakan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023/369
Record Dates: First submitted 2024-11-07; First posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-06

CONDITIONS: Caregiver Burnout; Caregiver; Care Burden
MeSH Terms: conditions — Caregiver Burden | interventions — Relaxin

STUDY DESIGN:
Intervention Model Description: Individuals assigned as intervention and control will complete the research in these groups.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention (Experimental)
  Interventions: Behavioral: relaxin
- control (Other)
  Interventions: Other: kontrol

INTERVENTIONS:
Behavioral: relaxin — caregivers relaxing and care burden
  Arms: intervention
Other: kontrol — no intervention
  Arms: control

SUMMARY:
Caregivers are also faced with multiple stress factors. Autogenic relaxation therapy will help caregivers relax and take time for themselves by getting away from the stressful life they have lived. Although there are various studies on this subject (Chegeni et al. 2018, Seo and Kim 2019, Ramiraz-Garcia et al. 2020, Wang et al. 2021, Bagheri et all 2021, Ozhanlı and Akyuz 2022), there is no study on caregivers as far as we could reach. As a result of this study, nurses will help caregivers, whom they work one-on-one in most areas, to relax, thus helping to increase the quality of patient care in home environments and contributing to the increase in the quality of life of the caregiver. Thus, caregivers will be able to manage care more actively and effectively both at home and in clinics.

Based on this purpose, the aim of the study is to reduce the anxiety level of caregivers, increase the quality of life and reduce the burden of care after autogenic relaxation therapy to be applied to caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old
* Being able to answer data collection forms
* Being able to speak Turkish
* Being able to provide continuous or partial care to a patient for at least 3 months
* Being able to communicate

Exclusion Criteria:

* Having epilepsy
* Not speaking or understanding Turkish
* Having a neurological disability
* Having had an acute myocardial infarction
* Being diagnosed with schizophrenia and major depression
* Being addicted to alcohol or drugs
* Having a history of loss of consciousness

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 64 (Estimated)
Dates: Start 2024-11-07 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-02-20 (Estimated)

PRIMARY OUTCOMES:
Principial | 1 month
  A decrease in the perceived stress scale score indicates a decrease in stress, an increase in the quality of life scale score indicates an increase in the quality of life, and a decrease in the care burden scale score indicates a decrease in the care burden. The secondary outcome measure is the decrease in the Perceived Stress Scale score, the increase in the Quality of Life Scale Score, and the decrease in the care burden scale score after autogenic relaxation therapy applied to caregivers.

SECONDARY OUTCOMES:
second | 3 month
  The secondary outcome measure is that caregivers feel better after autogenic relaxation therapy, are able to perform autogenic relaxation therapy on their own, and are least affected by the disadvantages of the care burden.

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan Üniversitesi, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No